CLINICAL TRIAL: NCT00341432
Title: Nicotine Replacement Therapy Methods for Pregnant Women
Brief Title: Effectiveness of Nicotine Replacement Therapy in Reducing the Risk of Nicotine Exposure in Pregnant Minority Smokers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 999905227; 05-CH-N227
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-04-20

CONDITIONS: Smoking; Pregnancy
Keywords: NRT Study; Smoking Cessation
MeSH Terms: conditions — Smoking; Smoking Cessation | interventions — Nicotine Replacement Therapy

INTERVENTIONS:
Behavioral: Nicotine Replacement Therapy

SUMMARY:
This study will compare the effectiveness of counseling plus use of a nicotine patch with counseling alone for helping pregnant women quit smoking. Smoking during pregnancy is the most preventable cause of fetal and newborn health problems such as low birth weight, fetal growth retardation, sudden infant death syndrome, spontaneous abortion, decreased lung function and premature delivery.

African-American and Hispanic women 18 years of age or older, smoke cigarettes, and live in the District of Columbia metropolitan area may be eligible for this study. Candidates are recruited from the George Washington University and Providence Hospital prenatal health clinics. They are screened with a review of their medical records and a survey that includes questions about their age, residency, race and ethnicity, educational level and employment status, number of weeks pregnant, and exposure to cigarette smoke and other types of tobacco.

Participants answer questions about their smoking behavior, then receive a 10-minute counseling session and watch a videotape about quitting smoking. Women who are not able to quit smoking in 1 week are then randomly assigned to one of two treatment groups. One group continues to receive counseling sessions during the remainder of their pregnancy; the second group receives nicotine patches as well as the counseling sessions. In addition, all participants watch a video about smoking and receive a guide to help them quit. Women who receive the patches must stop smoking completely. If they cannot stop immediately, their participation in the study ends. The behavioral counseling sessions for all the women are a series of conversations between the women and a trained counselor to help the woman through the process of quitting.

Participants are followed during the study with six clinic visits and three telephone calls. During the first visit, the women answer a series of questions about their smoking habits and health concerns. A portion of the urine sample they provide during their routine prenatal visit is used by this study to assess their cotinine (a breakdown product of nicotine) levels. Saliva and breath samples to test for cotinine and carbon monoxide levels are collected at each visit. Saliva is collected by brushing the inside of the cheek with a cotton swab, and breath samples are collected by having the woman blow into a tube connected to a machine. Participants are evaluated four times during the study with questions about their smoking behavior.

With the women's permission, their medical records, health, and treatments during pregnancy are reviewed. At the end of the pregnancy, the infant's weight and health are also reviewed.

DETAILED DESCRIPTION:
The overall focus of the proposed concept submitted by the George Washington University Medical Center investigators is "The Efficacy of NRT to Reduce the Risk of Nicotine Exposure in Pregnant Minority Smokers." Prenatal smoke exposure to the fetus and environmental tobacco smoke exposure of infants and children causes significant harm in both the short- and long-term. Smoking during pregnancy is the foremost preventable cause of perinatal morbidity and mortality. There is strong evidence that these exposures are associated with low birth weight (LBW) and infant mortality, respiratory illness, ear infections, tonsillectomy and adenoidectomy, asthma, and sudden infant death syndrome (SIDS), developmental delay, and increased health care utilization and hospitalizations.

George Washington University Medical Center investigators are submitting two concept papers that aim to test the efficacy of innovative intervention methods tailored to reduce fetal and infant exposure to nicotine secondary to maternal smoking and environmental tobacco exposure.

ELIGIBILITY:
* INCLUSION CRITERIA

At least 18 years of age

Resident of the District of Columbia or Greater Metropolitan Area

Minority Woman (Either African American or Hispanic)

No more than 30 weeks estimated gestational age

Able to read and speak English

Current cigarette smoker

Baseline saliva continine level equal to or exceeding 30 ng/ml

Expresses desire to quit smoking in this pregnancy

EXCLUSION CRITERIA

Currently participating in any other smoking cessation treatment program

Has the following conditions: heart disease, irregular heart beat, high blood pressure, diabetes, liver condition, kidney condition, stomach ulcer, asthma, chronic pulmonary disease, or skin condition

Currently being treated for psychiatric illness, alcoholism, or other drug addiction.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2005-08-16; Study Completion 2011-04-20 (Actual)

PRIMARY OUTCOMES:
Cotinine validated quit rates.

SECONDARY OUTCOMES:
Contine validated significant reduction.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - GW University Medical Center, Washington D.C., District of Columbia
  - Providence Hospital, Washington D.C., District of Columbia

REFERENCES:
- [Background] Mathews TJ, Menacker F, MacDorman MF. Infant mortality statistics from the 2000 period linked birth/infant death data set. Natl Vital Stat Rep. 2002 Aug 28;50(12):1-28. PMID 12224408
- [Background] Castles A, Adams EK, Melvin CL, Kelsch C, Boulton ML. Effects of smoking during pregnancy. Five meta-analyses. Am J Prev Med. 1999 Apr;16(3):208-15. doi: 10.1016/s0749-3797(98)00089-0. PMID 10198660
- [Background] Kleinman JC, Pierre MB Jr, Madans JH, Land GH, Schramm WF. The effects of maternal smoking on fetal and infant mortality. Am J Epidemiol. 1988 Feb;127(2):274-82. doi: 10.1093/oxfordjournals.aje.a114803. PMID 3337083
- [Derived] El-Mohandes AA, Windsor R, Tan S, Perry DC, Gantz MG, Kiely M. A randomized clinical trial of trans-dermal nicotine replacement in pregnant African-American smokers. Matern Child Health J. 2013 Jul;17(5):897-906. doi: 10.1007/s10995-012-1069-9. PMID 22761006
- [Derived] Tan S, Courtney LP, El-Mohandes AA, Gantz MG, Blake SM, Thornberry J, El-Khorazaty MN, Perry D, Kiely M. Relationships between self-reported smoking, household environmental tobacco smoke exposure and depressive symptoms in a pregnant minority population. Matern Child Health J. 2011 Dec;15 Suppl 1:S65-74. doi: 10.1007/s10995-011-0876-8. PMID 21928117